CLINICAL TRIAL: NCT03891693
Title: Biomimetic (SUPERA) Stent and Drug Eluting Balloon (Passeo 18 Lux) to Treat Recurrent Cephalic Arch Stenosis
Brief Title: Biomimetic Stent and Drug Eluting Balloon to Treat Recurrent Cephalic Arch Stenosis
Acronym: Arch-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2557
Record Dates: First submitted 2019-03-04; First posted 2019-03-27 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Brachiocephalic Vein Stenosis
Keywords: Stenosis; Angioplasty; Vascular Disease
MeSH Terms: conditions — Constriction, Pathologic; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: All subjects will be treated with SUPERA® stents and Passeo-18-Lux
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Passeo-18 Lux and SUPERA® stent (Experimental): Target lesion will be treated with Passeo-18 Lux Drug Eluting Balloon and SUPERA® stent during angioplasty
  Interventions: Device: Passeo-18 Lux and SUPERA® stent

INTERVENTIONS:
Device: Passeo-18 Lux and SUPERA® stent — Angioplasty of Arteriovenous Fistula (AVF) performed using Passeo-18 Lux and SUPERA® stent for patients with cephalic arch stenosis

SUMMARY:
The study evaluates the use of a biomimetic stent (SUPERA®) and a drug eluting balloon (DEB - Passeo 18 Lux) for the treatment of recurrent and tight cephalic arch stenosis in patients with brachiocephalic fistulas. All participants will undergo angioplasty with stated devices, and be followed up with over 12 months.

DETAILED DESCRIPTION:
To date, the treatment options are limited for recurrent and tight cephalic arch stenosis in patients with brachiocephalic fistulas - Angioplasty, with or without the placement of a stent, surgical bypass using the internal jugular vein or a cephalic/brachial venous anastomosis, or the creation of a new fistula may be a reasonable option. Angioplasty may be associated with technical failure and rupture of the arch vein in reported incidences of 24% and 6%, respectively. Percutaneous Transluminal Angioplasty (PTA) is associated with very low primary patency rates of 42% and 23% at 6 and 12 months, whilst bare stents are equally poor, with reported patency of 39% and 0% at those same time-point. The use of a biomimetic stent (SUPERA®) in the cephalic arch has not been studied to date, but may not only offer protection from rupture of the arch vein but may also create a material barrier to prevent the development of Neo-Intimal Hyperplasia (NIH). With the additional use of drug elution, this may impede NIH effect even more.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age is above 21 and below 90
* Informed consent obtained
* Chronic background treatment with daily ASA
* Patients with significant Cephalic Arch Vein Stenosis or recurrent stenosis within 6 months of initial POBA diagnosed either clinically or with Duplex Ultrasound
* Post-angioplasty cephalic arch lumen size between 5mm - 7mm maximum diameter

Exclusion Criteria:

* Patients with significant central vein stenosis (>70%) or total occlusion at time of angiographic study
* Cephalic arch stenosis <50% stenosis or diameter >5mm
* Patients with previous cephalic arch stenting (Bare Metal Stents or stent graft)
* Concomitant fistula inflow problem (e.g. juxta-anastomotic) that cannot be corrected optimally during the intervention (>30% residual stenosis or angiographic lumen <3mm)
* Patients with minor or major cephalic arch rupture during POBA procedure and the rupture point cannot be adequately sealed off during the procedure requiring a covered stent or open conversion
* Cephalic arch lesion length <10mm or greater than 10cm
* Patients with uncontrolled hypertension
* Patient <21 or > 90 years of age.
* Pregnant women or women of childbearing potential who are not following an effective method of contraception.
* Contraindication to aspirin or clopidogrel usage
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences o the study, or language barrier such that the subject is unable to give informed consent.
* Uncooperative attitude or potential for non-compliance with the requirements of the protocol making study participation impractical
* Patients who do NOT have impaired renal function
* Occluded or thrombosed fistula
* Patients presenting with central venous stenosis
* Final angioplasty treatment requires a stent or DEB >7mm in diameter
* Multiple lesions in the access circuit that cannot be treated with one stent and DEB.
* Vascular access circuit placed in the lower extremities
* Bare metal stent or stent-graft placed previously
* Metastatic caner or terminal medical condition
* Blood coagulation disorder
* Limited life expectancy (<6 months)
* Sepsis or active infection
* Recent arm thrombophlebitis
* Allergy or other known contraindication to iodinated media contrast, heparin or paclitaxel

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Angiographic Success | Immediately post-operation
  <30% regional stenosis within the stent and minimal lumen size should reach 5mm
Functional Fistula | Post-operation 1 week, 2 months, 6 months and 12 months.
  At the following time points, to monitor for any changes in whether fistula can be used successfully for dialysis without the need for re-intervention.
Primary Patency of Cephalic Arch | 1 year post-operation
  Less than 50% stenosis observed on duplex ultrasound

SECONDARY OUTCOMES:
Access Circuit Thrombosis | 1 year post-operation
  Thrombosis of access circuit requiring further intervention such as thrombolysis
Number of re-interventions per year | 1 year post-operation
  To note any re-interventions performed post-study procedure
Access Circuit Restenosis / Stent Fractures | 1 year post-operation
  To note any restenosis or stent fractures during study period that requires re-intervention
Access Circuit Infection | 1 year post-operation
  To note any infection at treated fistula during study period
Need for bypass revision surgery | 1 year post-operation

CONTACTS AND LOCATIONS:
Overall Officials: Tang Tjun Yip, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scheinert D, Werner M, Scheinert S, Paetzold A, Banning-Eichenseer U, Piorkowski M, Ulrich M, Bausback Y, Braunlich S, Schmidt A. Treatment of complex atherosclerotic popliteal artery disease with a new self-expanding interwoven nitinol stent: 12-month results of the Leipzig SUPERA popliteal artery stent registry. JACC Cardiovasc Interv. 2013 Jan;6(1):65-71. doi: 10.1016/j.jcin.2012.09.011. PMID 23347863
- [Background] Garcia L, Jaff MR, Metzger C, Sedillo G, Pershad A, Zidar F, Patlola R, Wilkins RG, Espinoza A, Iskander A, Khammar GS, Khatib Y, Beasley R, Makam S, Kovach R, Kamat S, Leon LR Jr, Eaves WB, Popma JJ, Mauri L, Donohoe D, Base CC, Rosenfield K; SUPERB Trial Investigators. Wire-Interwoven Nitinol Stent Outcome in the Superficial Femoral and Proximal Popliteal Arteries: Twelve-Month Results of the SUPERB Trial. Circ Cardiovasc Interv. 2015 May;8(5):e000937. doi: 10.1161/CIRCINTERVENTIONS.113.000937. PMID 25969545
- [Background] Bishu K, Armstrong EJ. Supera self-expanding stents for endovascular treatment of femoropopliteal disease: a review of the clinical evidence. Vasc Health Risk Manag. 2015 Jul 13;11:387-95. doi: 10.2147/VHRM.S70229. eCollection 2015. PMID 26203255
- [Background] Micari A, Brodmann M, Keirse K, Peeters P, Tepe G, Frost M, Wang H, Zeller T; IN.PACT Global Study Investigators. Drug-Coated Balloon Treatment of Femoropopliteal Lesions for Patients With Intermittent Claudication and Ischemic Rest Pain: 2-Year Results From the IN.PACT Global Study. JACC Cardiovasc Interv. 2018 May 28;11(10):945-953. doi: 10.1016/j.jcin.2018.02.019. PMID 29798770
- [Background] Zeller T, Beschorner U, Pilger E, Bosiers M, Deloose K, Peeters P, Scheinert D, Schulte KL, Rastan A, Brodmann M. Paclitaxel-Coated Balloon in Infrapopliteal Arteries: 12-Month Results From the BIOLUX P-II Randomized Trial (BIOTRONIK'S-First in Man study of the Passeo-18 LUX drug releasing PTA Balloon Catheter vs. the uncoated Passeo-18 PTA balloon catheter in subjects requiring revascularization of infrapopliteal arteries). JACC Cardiovasc Interv. 2015 Oct;8(12):1614-22. doi: 10.1016/j.jcin.2015.07.011. PMID 26493253
- [Background] Zhang D, Yang R, Wang S, Dong Z. Paclitaxel: new uses for an old drug. Drug Des Devel Ther. 2014 Feb 20;8:279-84. doi: 10.2147/DDDT.S56801. eCollection 2014. PMID 24591817
- [Background] Cho SB, Choi HC, Bae E, Park TJ, Baek HJ, Park SE, Ryu KH, Moon JI, Choi BH, Bae K, Jeon KN. Angioplasty and stenting for the proximal anastomotic stenosis of a brachio-axillary bypass graft using a helical interwoven nitinol stent: A case report. Medicine (Baltimore). 2017 Dec;96(50):e9073. doi: 10.1097/MD.0000000000009073. PMID 29390303
- [Derived] Tang TY, Tan CS, Yap C, Tan RY, Tay HH, Choke E, Chong TT. Helical stent (SUPERA) and drug-coated balloon (Passeo-18 Lux) for recurrent cephalic arch stenosis: Rationale and design of arch V SUPERA-LUX Study. J Vasc Access. 2020 Jul;21(4):504-510. doi: 10.1177/1129729819881589. Epub 2019 Oct 17. PMID 31621477